CLINICAL TRIAL: NCT03038048
Title: Intravitreal Injection Using 33-gauge Versus 30-gauge Needles: Comparison of Patients' Experience
Brief Title: 30g vs 33g Needle for Intravitreal Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, MidAtlantic Retina, Allen Chiang, MD, Wills Eye
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 16-594E
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Age Related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Degeneration; Retinal Vein Occlusion | interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 33 g needle - right eye (Experimental): 33 g needle for intravitreal injection of Lucentis or Eylea for right eye and 30 g needle for left eye
  Interventions: Procedure: Varying needle size with intravitreal ranibizumab or aflibercept
- 33 g needle - left eye (Experimental): 33 g needle for intravitreal injection of Lucentis or Eylea for left eye and 30 g needle for right eye
  Interventions: Procedure: Varying needle size with intravitreal ranibizumab or aflibercept

INTERVENTIONS:
Procedure: Varying needle size with intravitreal ranibizumab or aflibercept — Varying gauge of needle, 33 gauge vs 30 gauge
  Other Names: Lucentis, Eylea

SUMMARY:
We are comparing the patient experience between the standard 30 g needle to the smaller 33 g needle for intravitreal injections of ranabizumab or aflibercept for age related macular degeneration, diabetic macular edema, or retina vein occlusions.

DETAILED DESCRIPTION:
This is a prospective, randomized, interventional pilot study, which seeks to compare the patient experience using 30-gauge versus 33-gauge needle for bilateral same-day intravitreal injections of ranibizumab or aflibercept for the treatment of wet age-related macular degeneration (AMD), diabetic macular edema (DME), or macular edema associated with retinal vein occlusion (RVO). The null hypothesis is that there is no difference in patient discomfort or pain with the 30-gauge needle compared to the 33-gauge needle.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing bilateral, same-day, intravitreal injections of either ranibizumab oraflibercept for the diagnosis of wet AMD, DME, or RVO-associated macular edema

Exclusion Criteria:

* 1) Patients who do not receive Betadine ophthalmic solution prior to intravitreal injection due to documented allergy 2) Patients who are receiving intravitreal bevacizumab (this medication iscompounded into pre-filled 1-mL tuberculin syringes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Difference in discomfort between 30g and 33g needle | Day 1
  Intravitreal injection study pain questionnaire to evaluate discomfort associated with intravitreal injections

SECONDARY OUTCOMES:
Intraocular pressure 5 minutes post injection | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Allen Chiang, MD, Principal Investigator — Mid Atlantic Retina
Locations (1):
- Mid Atlantic Retina- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No